CLINICAL TRIAL: NCT03185871
Title: Celecoxib Window of Opportunity Trial to Assess Tumor and Stroma Responses
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UW16141; P30CA014520 (NIH); 2017-0219 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*H (Other: UW Madison)
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2018-10

CONDITIONS: Breast Carcinoma
Keywords: Invasive breast carcinoma; breast carcinoma stage T1cN0 to N3N0
MeSH Terms: conditions — Breast Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Masking Description: Due to the characteristics of the design of this clinical trial, the patient will not be blinded but the researcher completing analysis will be. The researcher will be handling deidentified patient samples and comparing whether there are changes of biological markers within the same patient before and after celecoxib intake. It is important that the researcher be as unbiased as possible when analyzing collagen alignment and amount of other breast cancer biological markers.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Celecoxib (Experimental): The participants will be scheduled for the two quantitative breast MRI exams. Following the first MRI exam, participants will start taking celecoxib 200mg twice a day with food. Subjects will take a minimum of 26 doses and no more than 32 doses of celecoxib during the study.
  Participants will intake 200mg of celecoxib two times a day (400mg/day total) for 2 weeks after biopsy. Histologic tissue samples will be obtained for evaluation at time of biopsy of the tumor and at time of surgery removal of the tumor.
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib — Celecoxib is the only COX-2 inhibitor currently approved by the FDA to be used in the United States. Recently, it has been shown that celecoxib prevents sporadic colorectal adenomas and there are more clinical trials evaluating the use of celecoxib in combination with chemotherapy regimens in breast cancer settings. Celebrex® oral capsules that will be used in this study contain 200 mg of celecoxib, in combination with inactive ingredients that include the following components: croscarmellose sodium, edible inks, gelatin, lactose monohydrate, magnesium stearate, povidone and sodium lauryl sulfate.
  Other Names: Celebrex

SUMMARY:
The overall purpose of this study is to assess whether celecoxib can reduce the change in collagen alignment and inflammatory response in the tumor tissue of primary breast cancer patients with invasive breast carcinoma after 2 weeks of oral intake.

DETAILED DESCRIPTION:
Advances in early detection techniques and improvement in systemic treatment of early stage breast cancer have led to a small decline in overall breast cancer mortality in the last 20 years. New advances will require understanding of breast cancer biology at the molecular level. Inhibition of COX-2 and its analysis of effect in breast cancer tumor microenvironment provide one such fruitful therapeutic target. Tumor microenvironment is poorly understood in breast cancer research. Despite new drugs being developed to treat breast cancer and tested in clinical trials, it is rarely possible to assess how the drug is affecting the breast cancer cells at a molecular level. The use of collagen properties such as alignment and deposition will allow giving a faster diagnosis of breast cancer status and seeing how celecoxib with respect to collagen can change the tumor microenvironment in human tissue. This window trial provides a way to look at cancer and stromal cells before and after celecoxib intake to see if the drug is actively working. If we can do this before and after a patient has surgery, and see how the tumor microenvironment responds, then the physician could pick a better suited adjuvant treatment for this patient after surgical intervention that would improve their overall survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have biopsy proven invasive breast carcinoma stages T1cN0 to T3N0, ER or PR positive with tumors greater than 1cm without lymph node spread.
* Participants must have a mammographic breast composition category (density) of c or d.
* Participants must be willing to participate and provide signed informed consent.
* Participants must have no immediate requirements for chemotherapy, radiotherapy or hormonal therapy.
* Participants must be willing to discontinue any use of NSAIDs like aspirin or ibuprofen until the tumor is removed
* Participants cannot be taking the following medications because of major pharmacokinetic interactions with celecoxib while being enrolled in the study: Abciximab, Argatroban, Bivalirudin, Cilostazol, Dabigatran, Etexilate, Dipyridamole, Fondaparinux, Heparin, Lepirudin, Pemetrexed, Protein C, Rivaroxaban, Sibutramine, Ticlopidine, Tirofiban, Vilazodone and Warfarin.
* Participants should pass MRI screening questionnaire

Exclusion Criteria:

* Prior history of cancer, neo-adjuvant chemotherapy and radiation therapy
* No daily NSAIDs intake within the past 4 weeks. Intermittent non-daily NSAIDs is allowed under PI discretion.
* Current or prior systemic use of corticosteroids in the past month.
* Participants with history of hypertension, congestive heart failure, edema, stroke or other cardiac disease or condition.
* Participants with type 2 diabetes, documented stomach ulcers and pulmonary embolism.
* Participants with aspirin or other NSAIDs-induced asthma or hypersensitivity reaction, sulfonamide allergy
* Participants who are currently pregnant
* Participants with known human immunodeficiency virus (HIV) infection, hepatitis B carrier state or with clinical evidence of hepatitis B.
* Participants who are not able to understand or provide written informed consent.
* Participants with standard contraindications to non-contrast MRI will be excluded, including claustrophobia and metallic implants incompatible with MRI.
* Participants whose girth exceeds the bore of the MRI scanner.
* Participants requiring conscious sedation for MR imaging.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Changes in collagen | Up to 6 weeks
  To determine change of collagen structure and proliferation in response to celecoxib intake in the tumor microenvironment.

SECONDARY OUTCOMES:
Change in correlation of collagen alignment and COX-2 expression | Up to 6 weeks
  To evaluate correlation among collagen alignment and COX-2 expression before and after celecoxib intake.
Changes in Syndecan-1 | Up to 6 weeks
  To analyze Syndecan-1 expression levels as stromal response biomarkers.
Changes in CD68 | Up to 6 weeks
  To analyze CD68 expression levels as stromal response biomarkers.
Changes in CD163 | Up to 6 weeks
  To analyze CD163 expression levels as stromal response biomarkers.
Changes in neutrophil elastase | Up to 6 weeks
  To analyze neutrophil elastase expression levels as stromal response biomarkers.
Changes in vimentin | Up to 6 weeks
  To analyze vimentin expression levels as stromal response biomarkers.
Changes in α-SMA | Up to 6 weeks
  To analyze α-SMA expression levels as stromal response biomarkers.
Changes in Ki67 | Up to 6 weeks
  To analyze Ki67 expression levels as stromal response biomarkers.
Changes in tissue cytokines in dense breast tissue | Up to 6 weeks
  To discover tissue cytokines present in dense breast tissue that are altered in response to celecoxib.
Number of subjects with adverse events associated with celecoxib | Up to 6 weeks
  To evaluate any adverse events associated with the 2-week intake of 200mg celecoxib twice a day.
Changes in collagen due to relationship of amount/percentage of fibroglandular tissue | Up to 6 weeks
  To determine if changes in collagen structure and proliferation in response to celecoxib differ by the amount and/or percentage of fibroglandular tissue, measured quantitatively using MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Burkard, MD, Principal Investigator — University of Wisconsin, Madison

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center Homepage — https://cancer.wisc.edu/